CLINICAL TRIAL: NCT00471237
Title: Study CR9108963: A 12-month, Randomized, Double-blind, Parallel-group, Placebo and Active-controlled Dose-range Finding Study of the Efficacy and Safety of SB-751689 in Post-menopausal Women With Osteoporosis
Brief Title: A Phase II Study Evaluating SB-751689 in Post-Menopausal Women With Osteoporosis.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated for futility by sponsor after a pre-planned interim review of data
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR9108963
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-09

CONDITIONS: Osteoporosis
Keywords: bone mineral density,; Ronacaleret; teriparatide; alendronate,; Post-menopausal women,; osteoporosis,; SB-751689
MeSH Terms: conditions — Osteoporosis | interventions — ronacaleret; Teriparatide; Alendronate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (No Intervention): All subjects will take calcium (500-660mg elemental daily) and vitamin D (at least 400IU daily) supplements once daily in the evening throughout the study
- Alendronate (Active Comparator): All subjects will take calcium (500-660mg elemental daily) and vitamin D (at least 400IU daily) supplements once daily in the evening throughout the study
  Interventions: Drug: Alendronate
- Teriparatide (Active Comparator): Open-label arm. All subjects will take calcium (500-660mg elemental daily) and vitamin D (at least 400IU daily) supplements once daily in the evening throughout the study
  Interventions: Drug: Teriparatide
- Ronacaleret (Experimental): 4 arms, 100mg, 200mg, 300mg, 400mg. All subjects will take calcium (500-660mg elemental daily) and vitamin D (at least 400IU daily) supplements once daily in the evening throughout the study.
  Interventions: Drug: Ronacaleret

INTERVENTIONS:
Drug: Ronacaleret — 100mg, 200mg, 300mg, 400mg
  Other Names: SB-751689
  Arms: Ronacaleret
Drug: Teriparatide — PTH (1-34)
  Arms: Teriparatide
Drug: Alendronate — Bisphosphonate
  Arms: Alendronate

SUMMARY:
This is a 12 month study designed to evaluate the safety and effectiveness of SB-751689 in the treatment of osteoporosis in post-menopausal women, in comparison with 2 active comparators and placebo.

ELIGIBILITY:
Inclusion:

* Informed consent: Subject is willing and able to provide written informed consent.
* Menopausal status: Ambulatory female aged < 80 years at screening and >5 years postmenopausal.
* T-Score: A subject with either no or only one prevalent vertebral fracture is eligible for inclusion if she satisfies one of the following T-score requirements:

If no prevalent vertebral fracture subject must have an absolute BMD value consistent with a T-score of less than or equal to -2.5 and greater than -4.0 at either the femoral neck, total hip, trochanter, or lumbar spine, or If one prevalent vertebral fracture subject must have an absolute BMD value consistent with a T-score of less than or equal to -2.0 and greater than -4.0 at either the femoral neck, total hip, trochanter, or lumbar spine.

* Suitable vertebra: Two or more vertebra in the range of L1 to L4 that are suitable for BMD measurement by DXA.
* Protocol compliance: Subject who, in the opinion of the investigator, is willing and able to comply with the requirements of the protocol.

Exclusion:

* T-Score: Has an absolute BMD value consistent with a T-score less than or equal to -4.0 at either the femoral neck, total hip, trochanter, or lumbar spine.
* Vertebral fractures: Has >1 prevalent vertebral fracture at the screening visit.
* Non-vertebral fractures: Any previous non-vertebral osteoporosis related/fragility fracture after age 40.
* Spine deformity: Significant spine deformity which would preclude DXA/QCT assessments.
* BMI: BMI ≥33kg/m2.
* Bone metabolic diseases: Other than osteoporosis, history or concurrent diseases affecting bone metabolism (e.g., osteomalacia, hyperparathyroidism, hyperthyroidism).
* GI disease: History of major upper gastrointestinal disease
* Malabsorption: Active or history of malabsorption (e.g., history of celiac disease, irritable bowel syndrome or inflammatory bowel disease).
* Liver disease: Past or current history of liver disease or known hepatic or biliary abnormalities, (with the exception of previously documented diagnosis of Gilbert's syndrome).
* Rheumatoid arthritis: Active disease or history of rheumatoid arthritis.
* Nephrolithiasis: History of or active nephrolithiasis (kidney stones).
* Osteosarcoma risk: Subjects at increased risk of osteosarcoma such as those with Paget's disease of bone or any prior external beam or implant radiation therapy involving the skeleton.
* Malignancy: Malignant disease diagnosed within the previous 5 years (except resected basal cell cancer).
* Biological abnormalities: Any clinically relevant biological abnormality found and/or volunteered at screening (other than those related to the disease under investigation) which, in the opinion of the investigator, is clinically significant and would preclude safe participation in this study.
* Surgical and medical conditions: Presence of the following conditions within six months prior to screening: myocardial infarction, coronary bypass surgery, coronary artery angioplasty, unstable angina, cardiac arrhythmia, clinically evident congestive heart failure, or cerebrovascular accident.
* Glomerular filtration rate: Glomerular filtration rate (GFR) <35 mL/min as calculated by the Modification of Diet in Renal Disease (MDRD) equation as follows: GFR (mL/min/1.73 m2) = 186 x (Serum creatinine mg/dL)-1.154 x (Age)-0.203 x (0.742 if female) x (1.210 if African American) (conventional units).
* QT/QTc prolongation: A marked baseline prolongation of QT/QTc interval (e.g., QTc interval ≥450 msec on the Screening ECG).
* Torsades de Pointes: A history of risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Liver chemistries: Liver chemistries [aspartate aminotransferase (AST), alanine aminotransferase (ALT) or total bilirubin] exceeding 2-fold the upper limit of the laboratory-specified reference range, at screening.
* Abnormal serum calcium: Serum calcium (total or albumin-adjusted) outside the central laboratory reference range at the screening visit.
* Abnormal PTH: PTH (intact or whole) outside the normal range.
* Abnormal creatine phosphokinase: Creatine phosphokinase (CPK) outside the normal range.
* Abnormal alkaline phosphatase: Alkaline phosphatase outside of the normal range.
* Thyroid hormone replacement: Subjects receiving thyroid hormone replacement therapy must have a TSH level checked. Subjects will be excluded if TSH levels are <0.1 or >10.0mIU/L. However, subjects will not be excluded if TSH is in the range 0.1-4.5 mIU/L. If TSH is >4.5 and ≤10.0mIU/mL, measure T4 and exclude the subject only if the T4 is outside the normal range.
* Vitamin D deficiency: Vitamin D deficiency (serum 25-hydroxy vitamin D < 20ng/mL, equivalent to 50nmol/L) at screening. Subjects can undergo vitamin D repletion as per local practice and be re-screened once only for vitamin D levels within the 6-week screening period. They will remain excluded if the re-screened value is < 20ng/mL.
* Previous strontium or IV bisphosphonate: Any previous treatment with strontium ranelate or intravenous bisphosphonate.
* Oral bisphosphonates: Any previous treatment with an oral bisphosphonate as follows:

any treatment within the last six months

* one month cumulative treatment within the last 12 months
* three months cumulative treatment within the past two years, or
* two years cumulative treatment within the past five years.

  * Fluoride: Treatment with fluoride (dose greater than 10mg/day) within the previous 5 years for osteoporosis.
  * Digoxin: Current therapy with digoxin.
  * Bone metabolism drugs: Treatment with other drugs affecting bone metabolism within the last six months prior to screening:

Chronic systemic corticosteroid [e.g., glucocorticoid, mineralocorticoid] treatment of no more than 2 intra-articular injections within the past year or use of oral, parenteral, or long-term, high-dose inhaled corticosteroids. Treatment with any topical corticosteroid will not exclude the subject from participating.

Hormones [e.g., estrogens/"natural estrogen preparations"(except for nonsystemic vaginal treatment), 19-norprogestins, SERMs such as raloxifene, anabolic steroids/androgens such as dehydroepiandrosterone (DHEA) or its sulfated form (DHEAS), nandrolone, tibolone, active vitamin D analogs/metabolites such as 1,25-dihydroxy vitamin D (calcitriol) or 1alpha-hydroxyvitamin D3 (1-alpha hydroxycholecalciferol), calcitonin].

Calcineurin inhibitors [e.g., cyclosporine, tacrolimus] or methotrexate.

* Previous anabolic agents: Treatment with PTH, PTH analogues or similar anabolic agent for osteoporosis within the last two years.
* Contraindications: Contraindications to therapy with calcium or vitamin D.
* Pregnancy: Women who are pregnant are not allowed in this study.
* Interfering medications: Vitamin A in excess of 10,000 IU per day, heparin, or lithium, or anticonvulsant medications except benzodiazepines.
* Investigational drug exposure: Administration of any investigational drug within 90 days preceding the first dose of the study drug.
* Substance abuse: History or current evidence of drug or alcohol abuse within the previous 12 months.
* Problems swallowing: Inability to swallow a tablet whole.

The following exclusion criteria do not apply to subjects allocated to the open-label teriparatide group:

* Calcium channel blockers: Current therapy with calcium channel blockers diltiazem and verapamil.
* Oral Azole Antifungals: Current therapy with any oral azole antifungal.
* Immunosuppressants: Current therapy with cyclosporine or oral tacrolimus.
* Ritonavir: Current therapy with ritonavir.
* Quinidine: Current therapy with quinidine.
* Macrolide Antibiotics: Subjects anticipated to require chronic use of macrolide antibiotics.
* Alendronate Contraindications: Contraindications to therapy with alendronate. Additional Exclusion Criteria for Subjects Recruited at QCT Sites
* Hip surgery: History of hip surgery resulting in a metal implant on either the left or right side that would cause an artefact on a QCT scan.

Additional Exclusion Criteria for Teriparatide Subjects

* Teriparatide contraindications: Contraindications to therapy with teriparatide according to locally approved datasheet.

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2007-05-14 (Actual); Primary Completion 2008-12-26 (Actual); Study Completion 2008-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (9):
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Palm Desert, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Duncansville, Pennsylvania
- Argentina (2):
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Australia (4):
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Footscray, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
- Belgium (3):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Tienen
- GSK Investigational Site, Ballerup Municipality, Denmark
- Germany (3):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hong Kong (2):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin
- GSK Investigational Site, Mexico City, Mexico
- Norway (3):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Oslo
- Poland (3):
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- GSK Investigational Site, Moscow, Russia
- South Africa (3):
  - GSK Investigational Site, Panorama
  - GSK Investigational Site, Rosebank
  - GSK Investigational Site, Somerset West
- South Korea (2):
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Fitzpatrick LA, Dabrowski CE, Cicconetti G, Gordon DN, Fuerst T, Engelke K, Genant HK. Ronacaleret, a calcium-sensing receptor antagonist, increases trabecular but not cortical bone in postmenopausal women. J Bone Miner Res. 2012 Feb;27(2):255-62. doi: 10.1002/jbmr.554. PMID 22052452
- [Derived] Fitzpatrick LA, Dabrowski CE, Cicconetti G, Gordon DN, Papapoulos S, Bone HG 3rd, Bilezikian JP. The effects of ronacaleret, a calcium-sensing receptor antagonist, on bone mineral density and biochemical markers of bone turnover in postmenopausal women with low bone mineral density. J Clin Endocrinol Metab. 2011 Aug;96(8):2441-9. doi: 10.1210/jc.2010-2855. Epub 2011 May 18. PMID 21593114
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: CR9108963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: CR9108963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: CR9108963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: CR9108963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: CR9108963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: CR9108963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: CR9108963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 14-May-2007and 26-December-2008 at 45 centres in 14 countries.
Pre-assignment Details: Of the 1609 participants screened, 1040 were screen failures, remaining 569 were randomized to the treatment arms. One participant from each of the 4 ronacaleret groups and alendronate group were excluded from Intent-to-Treat population and 564 participants were included in Intent-to-Treat population.
Groups:
- Placebo: Participants received matching placebo once daily (OD) (matching to ronacaleret tablet) and matching placebo once weekly (OW) (matching to Alendronate capsule) for 12 months. Participants were supplied with elemental calcium 500-660 milligrams (mg) and vitamin D, at least 400 international units (IU), OD in the evening as dietary supplements throughout the study.
- Ronacaleret, 100 mg Tablet, OD: Participants received ronacaleret, 100 mg tablet, OD and matching placebo, OW (matching to Alendronate capsule) for 12 months. Participants were supplied with elemental calcium 500-660 mg and vitamin D, at least 400 IU, OD in the evening as dietary supplements throughout the study.
- Ronacaleret, 200 mg Tablet, OD: Participants received ronacaleret, 200 mg tablet, OD and matching placebo, OW (matching to Alendronate capsule) for 12 months. Participants were supplied with elemental calcium 500-660 mg and vitamin D, at least 400 IU, OD in the evening as dietary supplements throughout the study.
- Ronacaleret, 300 mg Tablet, OD: Participants received ronacaleret, 300 mg tablet, OD and matching placebo, OW (matching to Alendronate capsule) for 12 months. Participants were supplied with elemental calcium 500-660 mg and vitamin D, at least 400 IU, OD in the evening as dietary supplements throughout the study.
- Ronacaleret, 400 mg Tablet, OD: Participants received Ronacaleret, 400 mg tablet, OD and matching placebo, OW (matching to Alendronate capsule) for 12 months. Participants were supplied with elemental calcium 500-660 mg and vitamin D, at least 400 IU, OD in the evening as dietary supplements throughout the study.
- Alendronate, 70 mg, Capsule, OW: Participants received Alendronate, 70 mg, capsule, OW and matching placebo OD (matching to ronacaleret tablet) for 12 months. Participants were supplied with elemental calcium 500-660 mg and vitamin D, at least 400 IU, OD in the evening as dietary supplements throughout the study.
- Teriparatide, 20 mcg, SC Injection, OD: Participants received Teriparatide, 20 microgram (mcg), subcutaneous (SC) injection, OD for 12 months. Participants were supplied with elemental calcium 500-660mg and vitamin D, at least 400 IU, OD in the evening as dietary supplements throughout the study.
Period: Overall Study
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Started | 90 | 87 | 82 | 88 | 87 | 89 | 41
Completed | 49 | 45 | 48 | 43 | 46 | 50 | 38
Not Completed | 41 | 42 | 34 | 45 | 41 | 39 | 3
Not completed — Adverse Event | 6 | 5 | 4 | 8 | 7 | 5 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 2 | 3 | 0 | 0
Not completed — Protocol Violation | 3 | 6 | 3 | 2 | 2 | 4 | 1
Not completed — Withdrawal by Subject | 8 | 6 | 5 | 8 | 7 | 4 | 2
Not completed — Sponsor terminated study | 20 | 23 | 19 | 22 | 18 | 24 | 0
Not completed — Non-compliance | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Met serum creatinine withdrawal criteria | 1 | 0 | 2 | 2 | 0 | 0 | 0
Not completed — Early stopping due to non-efficacy | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant planned to travel to abraod | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — High parathyroid hormone | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant lost medication | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Administration of prohibited medicine | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant shifted residence | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant's decision | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received matching placebo OD (matching to ronacaleret tablet) and matching placebo OW (matching to Alendronate capsule) for 12 months. Participants were supplied with elemental calcium 500-660 mg and vitamin D, at least 400 IU, OD in the evening as dietary supplements throughout the study.
- Teriparatide, 20 mcg, SC Injection, OD: Participants received Teriparatide, 20 mcg, SC injection, OD for 12 months. Participants were supplied with elemental calcium 500-660mg and vitamin D, at least 400 IU, OD in the evening as dietary supplements throughout the study.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD | Total
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41 | 564
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.20 (6.75) | 64.17 (7.69) | 64.16 (7.03) | 64.34 (6.57) | 64.97 (7.60) | 65.11 (7.04) | 63.17 (5.92) | 64.24 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 87 | 82 | 88 | 87 | 89 | 41 | 564
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participant]
  African American/African Heritage | 1 | 2 | 1 | 0 | 4 | 1 | 0 | 9
  American Indian or Alaska Native | 5 | 5 | 3 | 3 | 1 | 4 | 3 | 24
  Asian | 10 | 7 | 10 | 11 | 10 | 8 | 3 | 59
  White | 73 | 71 | 66 | 73 | 71 | 76 | 35 | 465
  African American/African Heritage & White | 1 | 2 | 2 | 1 | 1 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Bone Marrow Density (BMD) at Month 12 Measured by Dual-Energy X-Ray Absorptiometry (DXA) Scans of the Lumbar Spine (L1-L4)
Description: DXA scanners from Hologic and GE Lunar was used to measure BMD by a DXA scan. At least two vertebrae (L1-L4) that were suitable for measurement of BMD were evaluated. The same scanner was used throughout the study for all measurements for a given participant. DXA scans were sent to a central reading facility for quality control and central analysis. Assessments performed on Day 0 were considered as Baseline. Percent change from Baseline was computed as (change from baseline / baseline value) * 100%. Percent change from Baseline in areal bone mineral density (aBMD) was reported.
Time Frame: Baseline (Day 0) and 12 Months
Population: Intent-to-Treat population comprised of any randomised or teriparatide participant who received at least one dose of study medication. Only those participants available at the specified time points were analyzed. Teriparatide arm was excluded from the analysis, since these participants were not randomized and were disproportionately represented.
Measure: Least Squares Mean (Standard Error); unit: Percent change in BMD
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW
Number analyzed (Participants) | 79 | 76 | 74 | 78 | 72 | 75
Percent change in BMD | 0.03 (0.38) | 0.32 (0.40) | 1.39 (0.40) | 1.61 (0.39) | 1.62 (0.40) | 4.54 (0.40)
Statistical Analysis 1: Comparison: Placebo vs Ronacaleret, 100 mg Tablet, OD; Test type: Superiority; p = 0.590, ANOVA; Each dose of ronacaleret was deemed significantly different from placebo if the Hommel-adjusted p-value was <0.044 at Month 12; Mean Difference (Net) = 0.29, 95% CI 2-sided [-0.78 to 1.37], Standard Error of Mean 0.55
Statistical Analysis 2: Comparison: Placebo vs Ronacaleret, 200 mg Tablet, OD; Test type: Superiority; p = 0.028, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.36, 95% CI 2-sided [0.28 to 2.44], Standard Error of Mean 0.55
Statistical Analysis 3: Comparison: Placebo vs Ronacaleret, 300 mg Tablet, OD; Test type: Superiority; p = 0.011, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.58, 95% CI 2-sided [0.51 to 2.65], Standard Error of Mean 0.54
Statistical Analysis 4: Comparison: Placebo vs Ronacaleret, 400 mg Tablet, OD; Test type: Superiority; p = 0.012, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.60, 95% CI 2-sided [0.51 to 2.69], Standard Error of Mean 0.55

2. Primary Outcome: Number of Participants With Hypercalcemia
Description: Participants with albumin-adjusted serum calcium pre-dose values of >11.0 mg/ deciliter (dL) or post-dose values of >12.0 mg/dL were recorded as participants with hypercalcemia. Number of participant with hypercalcemia were reported.
Time Frame: Up to Month 12
Population: Intent-to-Treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41
Participants | 0 | 1 | 1 | 4 | 11 | 0 | 1

3. Primary Outcome: Number of Participants Withdrew Due to Hypercalcemia
Description: A confirmed albumin-adjusted serum calcium pre-dose value of >11.0 mg/dL or post-dose value of >12.0 mg/dL was set as a withdrawal criteria for the study. Number of participants who met this pre-defined stopping criteria were reported.
Time Frame: Up to Month 12
Population: Intent-to-Treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participant With Laboratory Abnormalities of Potential Clinical Concern at Any Post-baseline Visit
Description: The hematology parameters analyzed were white blood cells (WBC) count with differential WBC count, red blood cells, haemoglobin, haematocrit, mean corpuscular volume and platelet count. The clinical chemistry parameters analyzed were sodium, potassium, calcium, calcium (albumin adjusted), phosphate, bicarbonate, creatinine, bilirubin (total), alanine amino transferase, aspartate amino transferase, glucose, albumin, alkaline phosphatase, creatine phosphokinase, urea, uric acid, total protein, 25-OH vitamin D, 1,25-2(OH) vitamin D, whole parathyroid hormone (PTH 1-84)) and intact PTH (1-84 and 7-84). Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important laboratory findings at any visit were reported.
Time Frame: Up to Month 12
Population: Intent-to-Treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41
Participants
  Monocytes- high | 17 | 14 | 19 | 17 | 18 | 28 | 6
  Total neutrophils- high | 9 | 11 | 10 | 10 | 4 | 6 | 4
  Total neutrophils- low | 16 | 5 | 8 | 8 | 14 | 13 | 4
  Eosinophils- high | 12 | 8 | 11 | 18 | 19 | 11 | 6
  Glucose- high | 10 | 6 | 9 | 5 | 4 | 5 | 3
  Glucose- low | 3 | 0 | 4 | 0 | 3 | 0 | 0
  Basophils- high | 2 | 0 | 1 | 0 | 1 | 1 | 0
  Hematocrit- low | 2 | 0 | 0 | 2 | 0 | 0 | 1
  Hemoglobin- high | 1 | 0 | 1 | 0 | 1 | 0 | 1
  Hemoglobin- low | 2 | 0 | 0 | 2 | 1 | 0 | 1
  Platelets- high | 2 | 0 | 1 | 0 | 0 | 1 | 0
  White Blood Cell- high | 1 | 0 | 2 | 0 | 1 | 0 | 1
  White Blood Cell- low | 1 | 1 | 0 | 2 | 0 | 0 | 0
  Calcium- high | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Phosphorus- high | 1 | 0 | 0 | 1 | 0 | 0 | 1
  Alkaline Phosphatase- high | 0 | 1 | 0 | 3 | 3 | 1 | 0
  Total bilirubin- high | 0 | 1 | 2 | 1 | 1 | 0 | 0

5. Primary Outcome: Number of Participant With Vital Signs of Potential Clinical Concern at Any Post-baseline Visit
Description: The potential clinical importance ranges (low and high) of the vital sign parameters-systolic blood pressure (> 30 millimeter of mercury [mmHg] decrease from Baseline, > 30 mmHg increase from Baseline), diastolic blood pressure (> 20 mmHg decrease from Baseline and > 20 mmHg increase from Baseline) and heart rate (<45 and >120 beats per minute). Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important vital parameter findings at any visit were reported.
Time Frame: Up to 12 Months
Population: Intent-to-Treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41
Participants
  Systolic Blood Pressure, High: number analyzed (Participants) | 87 | 85 | 82 | 87 | 87 | 89 | 40
  Systolic Blood Pressure, High | 5 | 10 | 8 | 9 | 11 | 8 | 1
  Systolic Blood Pressure, Low: number analyzed (Participants) | 87 | 85 | 82 | 87 | 87 | 89 | 40
  Systolic Blood Pressure, Low | 6 | 8 | 10 | 6 | 4 | 8 | 3
  Diastolic Blood Pressure, High: number analyzed (Participants) | 87 | 85 | 82 | 87 | 87 | 89 | 40
  Diastolic Blood Pressure, High | 2 | 6 | 5 | 1 | 6 | 3 | 1
  Diastolic Blood Pressure, Low: number analyzed (Participants) | 87 | 85 | 82 | 87 | 87 | 89 | 40
  Diastolic Blood Pressure, Low | 8 | 9 | 4 | 12 | 10 | 10 | 2
  Heart Rate, Low: number analyzed (Participants) | 87 | 85 | 82 | 87 | 87 | 89 | 40
  Heart Rate, Low | 2 | 0 | 1 | 1 | 1 | 0 | 0

6. Primary Outcome: Number of Participant With Electrocardiogram (ECG) Findings Reported as Adverse Event
Description: Full 12-lead ECGs pre-dose at screening and visits 6, 8, 11, 12 and 14 were recorded. Participants rested supine or seated for at least 10 minutes before each reading. All ECGs were transmitted to a central reviewer for blinded assessment. The central reviewer measured the following parameters and provide a clinical interpretation: heart rate, RR interval, PR interval, QRS interval, QT (uncorrected) interval, QTcB (Bazett's correction) interval, QTcF (Fridericia's correction) interval. The central reviewer was provided the investigator or designated qualified site physician with a central ECG report or confirmatory report to assist them in identifying any clinically significant abnormalities that would preclude the participant from further participation in the study.
Time Frame: Up to 12 months
Population: Intent-to-Treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41
Participants | 1 | 5 | 4 | 3 | 3 | 5 | 0

7. Primary Outcome: Mean Change From Baseline in Height
Description: Assessments performed on Day 0 were considered as Baseline. Change from Baseline was computed as values at post baseline visit minus Baseline value. Mean change from baseline in height at Month 6 and 12 and early withdrawal were reported.
Time Frame: Baseline (Day 0), Month 6, 12 and early withdrawal
Population: Intent-to-Treat population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41
Centimeter
  Month 6: number analyzed (Participants) | 68 | 70 | 68 | 75 | 70 | 74 | 38
  Month 6 | -0.04 (0.58) | 0.17 (1.41) | 0.72 (3.82) | 0.05 (0.70) | -0.04 (0.82) | -0.07 (1.13) | 0.11 (0.65)
  Month 12: number analyzed (Participants) | 49 | 45 | 48 | 43 | 41 | 50 | 38
  Month 12 | -0.14 (0.65) | 0.04 (1.59) | 0.02 (0.76) | -0.09 (1.04) | -0.17 (0.67) | -0.08 (0.57) | 0.11 (0.56)
  Early withdrawal: number analyzed (Participants) | 36 | 36 | 32 | 37 | 31 | 35 | 2
  Early withdrawal | 0.03 (0.61) | 0.17 (1.92) | -0.13 (0.55) | -0.16 (0.76) | -0.16 (0.82) | -0.37 (0.88) | 0 (0)

8. Primary Outcome: Mean Change From Baseline in Weight
Description: Baseline values were assessed on Day 0. Change from Baseline was computed as values at post baseline visit minus Baseline value. Mean change from baseline in weight at Month 6, 12 and early withdrawal were reported.
Time Frame: Baseline (Day 0), Month 6, 12 and early withdrawal
Population: Intent-to-Treat population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41
Kilogram
  Month 6: number analyzed (Participants) | 69 | 70 | 68 | 75 | 70 | 74 | 38
  Month 6 | -0.02 (2.12) | 0.27 (3.27) | 0.45 (2.98) | -0.24 (2.87) | 0.11 (2.84) | 0.29 (1.89) | 0.51 (1.84)
  Month 12: number analyzed (Participants) | 49 | 45 | 48 | 43 | 47 | 50 | 38
  Month 12 | 0.32 (2.73) | -0.72 (2.70) | 1.18 (9.78) | -0.22 (2.36) | -0.48 (2.28) | 0.57 (3.22) | 0.09 (2.45)
  Early withdrawal: number analyzed (Participants) | 36 | 36 | 32 | 37 | 32 | 35 | 2
  Early withdrawal | -0.45 (2.40) | 0.40 (4.60) | -0.34 (2.48) | 0.37 (3.86) | 0.00 (2.17) | -0.12 (2.33) | -2.15 (1.48)

9. Secondary Outcome: Percent Change From Baseline to Month 6 in BMD Measured by DXA Scans of the Lumbar Spine (L1-L4)
Description: DXA scanners from Hologic and GE Lunar was used to measure BMD by a DXA scan. At least two vertebrae (L1-L4) that were suitable for measurement of BMD were evaluated. The same scanner was used throughout the study for all measurements for a given participant. DXA scans were sent to a central reading facility for quality control and central analysis. Baseline values were assessed on Day 0. Percent Change from Baseline was computed as (change from baseline / baseline value) * 100%. Percent change from baseline to month 6 in aBMD was reported.
Time Frame: Baseline (Day 0) and Month 6
Population: Intent to Treat Population. Only those participants available at the specified time point were analyzed. Participants from Teriparatide, 20 mcg, SC injection, OD arm were excluded from the analysis, since these participants were not randomized and were disproportionately represented.
Measure: Least Squares Mean (Standard Error); unit: percent change in BMD
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW
Number analyzed (Participants) | 79 | 76 | 74 | 77 | 73 | 75
percent change in BMD | 0.66 (0.33) | 0.21 (0.34) | 1.61 (0.35) | 0.47 (0.34) | 1.01 (0.35) | 3.42 (0.34)
Statistical Analysis 1: Comparison: Placebo vs Ronacaleret, 100 mg Tablet, OD; Test type: Superiority; p = 0.680, ANOVA; Each dose of ronacaleret was deemed significantly different from placebo if the Hommel-adjusted p-value was <0.006 at Month 6; Mean Difference (Net) = -0.45, 95% CI 2-sided [-1.38 to 0.48], Standard Error of Mean 0.47
Statistical Analysis 2: Comparison: Placebo vs Ronacaleret, 200 mg Tablet, OD; Test type: Superiority; p = 0.192, ANOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.95, 95% CI 2-sided [0.01 to 1.89], Standard Error of Mean 0.48
Statistical Analysis 3: Comparison: Placebo vs Ronacaleret, 300 mg Tablet, OD; Test type: Superiority; p = 0.680, ANOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.19, 95% CI 2-sided [-1.12 to 0.73], Standard Error of Mean 0.47
Statistical Analysis 4: Comparison: Placebo vs Ronacaleret, 400 mg Tablet, OD; Test type: Superiority; p = 0.680, ANOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.35, 95% CI 2-sided [-0.59 to 1.29], Standard Error of Mean 0.48

10. Secondary Outcome: Percent Change From Baseline to Months 6 and 12 in BMD Measured by DXA Scans of the Hip (Total Hip, Femoral Neck and Trochanter).
Description: DXA scanners from Hologic and GE Lunar was used to measure BMD by a DXA scan. At least two vertebrae (L1-L4) that were suitable for measurement of BMD were evaluated. The same scanner was used throughout the study for all measurements for a given participant. DXA scans were sent to a central reading facility for quality control and central analysis. Baseline values were assessed on Day 0. Percent Change from Baseline was computed as (change from baseline / baseline value) * 100%. Percent change from baseline to month 6 and 12 in aBMD of hip (total hip, femoral neck and trochanter) were reported.
Time Frame: Baseline (Day 0), Month 6 and Month 12
Population: Intent-to-Treat population. Only those participants available at the specified time points were analyzed. Participants from Teriparatide, 20 mcg, SC injection, OD arm were excluded from the analysis, since these participants were not randomized and were disproportionately represented.
Measure: Least Squares Mean (Standard Error); unit: Percent change in BMD
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89
Percent change in BMD
  Total Hip aBMD, Month 6: number analyzed (Participants) | 79 | 75 | 74 | 77 | 71 | 74
  Total Hip aBMD, Month 6 | 0.42 (0.23) | -0.26 (0.24) | -0.37 (0.24) | -0.86 (0.23) | -0.88 (0.24) | 1.84 (0.24)
  Total Hip aBMD, Month 12: number analyzed (Participants) | 79 | 75 | 74 | 78 | 70 | 74
  Total Hip aBMD, Month 12 | 0.27 (0.26) | -0.62 (0.26) | -0.75 (0.27) | -1.07 (0.26) | -1.31 (0.27) | 2.70 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Ronacaleret, 100 mg Tablet, OD; Total Hip aBMD, Month 6; Test type: Superiority; p = 0.037, ANOVA; Mean Difference (Net) = -0.68, 95% CI 2-sided [-1.32 to -0.04], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: Placebo vs Ronacaleret, 200 mg Tablet, OD; Total Hip aBMD, Month 6; Test type: Superiority; p = 0.017, ANOVA; Mean Difference (Net) = -0.79, 95% CI 2-sided [-1.43 to -0.14], Standard Error of Mean 0.33
Statistical Analysis 3: Comparison: Placebo vs Ronacaleret, 300 mg Tablet, OD; Total Hip aBMD, Month 6; Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Net) = -1.28, 95% CI 2-sided [-1.92 to -0.64], Standard Error of Mean 0.32
Statistical Analysis 4: Comparison: Placebo vs Ronacaleret, 400 mg Tablet, OD; Total Hip aBMD, Month 6; Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Net) = -1.30, 95% CI 2-sided [-1.95 to -0.65], Standard Error of Mean 0.33
Statistical Analysis 5: Comparison: Placebo vs Ronacaleret, 100 mg Tablet, OD; Total Hip aBMD, Month 12; Test type: Superiority; p = 0.015, ANOVA; Mean Difference (Net) = -0.89, 95% CI 2-sided [-1.61 to -0.17], Standard Error of Mean 0.36
Statistical Analysis 6: Comparison: Placebo vs Ronacaleret, 200 mg Tablet, OD; Total Hip aBMD, Month 12; Test type: Superiority; p = 0.006, ANOVA; Mean Difference (Net) = -1.02, 95% CI 2-sided [-1.74 to -0.30], Standard Error of Mean 0.37
Statistical Analysis 7: Comparison: Placebo vs Ronacaleret, 300 mg Tablet, OD; Total Hip aBMD, Month 12; Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Net) = -1.33, 95% CI 2-sided [-2.04 to -0.63], Standard Error of Mean 0.36
Statistical Analysis 8: Comparison: Placebo vs Ronacaleret, 400 mg Tablet, OD; Total Hip aBMD, Month 12; Test type: Superiority; p = 0.000, ANOVA; Median Difference (Net) = -1.57, 95% CI 2-sided [-2.30 to -0.84], Standard Error of Mean 0.37

11. Secondary Outcome: Number of Participants Who Remained the Same or Had Any Improvement in DXA BMD (> Baseline)
Description: Responder rate of participants who remained the same or had any improvement as compared to baseline in DXA BMD of vertebra, femur and vertebra plus femur were reported. Baseline values were assessed on Day 0. Percent change (improvement) from Baseline was computed as (change from baseline / baseline value) * 100%.
Time Frame: Baseline (Day 0), Month 5, 6 and 12
Population: Intent-to-Treat population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41
Participants
  Month 5, Vertebra, BMD % change >=0: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Month 5, Vertebra, BMD % change >=0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Month 5, Femur, BMD % change >=0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Month 5, Femur, BMD % change >=0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Month 5, Vertebra + Femur, BMD % change >=0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Month 5, Vertebra + Femur, BMD % change >=0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Month 6, Vertebra, BMD % change >=0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Month 6, Vertebra, BMD % change >=0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Month 6, Femur, BMD % change >=0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Month 6, Femur, BMD % change >=0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Month 6, Vertebra + Femur, BMD % change >=0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Month 6, Vertebra + Femur, BMD % change >=0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Month 12, Vertebra, BMD % change >=0: number analyzed (Participants) | 42 | 50 | 43 | 43 | 41 | 49 | 36
  Month 12, Vertebra, BMD % change >=0 | 16 | 29 | 32 | 35 | 31 | 44 | 34
  Month 12, Femur, BMD % change >=0: number analyzed (Participants) | 41 | 47 | 40 | 39 | 37 | 45 | 26
  Month 12, Femur, BMD % change >=0 | 20 | 23 | 14 | 19 | 16 | 40 | 25
  Month 12, Vertebra + Femur, BMD % change >=0: number analyzed (Participants) | 39 | 47 | 40 | 39 | 37 | 42 | 25
  Month 12, Vertebra + Femur, BMD % change >=0 | 10 | 19 | 12 | 17 | 16 | 35 | 24
  Early Withdrawal, Vertebra, BMD % change >=0: number analyzed (Participants) | 3 | 2 | 2 | 3 | 1 | 0 | 1
  Early Withdrawal, Vertebra, BMD % change >=0 | 1 | 1 | 1 | 2 | 1 | 0 | 1
  Early Withdrawal, Femur, BMD % change >=0: number analyzed (Participants) | 2 | 2 | 2 | 3 | 1 | 0 | 1
  Early Withdrawal, Femur, BMD % change >=0 | 1 | 1 | 0 | 1 | 1 | 0 | 1
  Early Withdrawal, Vertebra + Femur, BMD %change>=0: number analyzed (Participants) | 2 | 2 | 2 | 3 | 1 | 0 | 1
  Early Withdrawal, Vertebra + Femur, BMD %change>=0 | 1 | 1 | 0 | 1 | 1 | 0 | 1

12. Secondary Outcome: Percent Change From Baseline to Month 12 in the Volumetric Integral, Cortical, and Trabecular Density (BMD) at the Hip and Lumbar Spine as Measured by Quantitative Computer Tomography (QCT) Scans
Description: QCT is a three-dimensional non-projectional technique to quantify BMD with a number of advantages to other densitometric techniques. Cortical and trabecular bone can be separated, trabecular volume of interest (VOI) are largely independent of degenerative changes in the spine and 3 dimensional geometric parameters can be determined. BMD as measured by QCT is a true density measured in g/cm^3 in contrast to DXA Which determines an areal density measured in g/cm^2. Baseline values were assessed on Day 0. Percent change from Baseline was computed as (change from baseline / baseline value) * 100%. Percent change from Baseline to month 12 in the volumetric integral, cortical, and trabecular density (BMD) at the hip and lumbar spine measured by QCT were reported.
Time Frame: Baseline (Day 0) and Month 12
Population: Intent-to-Treat population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change in BMD
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41
Percent change in BMD
  Total vertebra integral VOI BMD: number analyzed (Participants) | 42 | 50 | 43 | 43 | 41 | 49 | 36
  Total vertebra integral VOI BMD | -0.98 (3.13) | 1.09 (4.01) | 3.00 (4.98) | 3.91 (4.98) | 4.83 (6.56) | 5.04 (4.39) | 14.80 (8.69)
  Mid vertebra integral VOI BMD: number analyzed (Participants) | 42 | 50 | 43 | 43 | 41 | 49 | 36
  Mid vertebra integral VOI BMD | -1.31 (3.54) | 1.20 (4.85) | 4.65 (5.87) | 6.06 (6.48) | 7.33 (8.67) | 4.85 (5.25) | 17.97 (11.27)
  Mid Cylinder trabecular VOI BMD: number analyzed (Participants) | 42 | 50 | 43 | 43 | 41 | 49 | 36
  Mid Cylinder trabecular VOI BMD | -2.45 (4.39) | 1.75 (8.70) | 6.17 (10.37) | 8.99 (10.52) | 13.29 (15.32) | 4.88 (7.68) | 24.37 (15.92)
  Mid Osteo trabecular VOI BMD: number analyzed (Participants) | 42 | 50 | 43 | 43 | 41 | 49 | 36
  Mid Osteo trabecular VOI BMD | -2.21 (4.58) | 1.81 (8.26) | 7.06 (9.25) | 9.54 (9.79) | 13.21 (14.68) | 5.15 (6.86) | 24.21 (15.80)
  Total vertebra trabecular VOI BMD: number analyzed (Participants) | 42 | 50 | 43 | 43 | 41 | 49 | 36
  Total vertebra trabecular VOI BMD | -2.46 (4.58) | 1.67 (7.18) | 5.81 (8.31) | 8.52 (8.97) | 11.40 (12.83) | 4.97 (6.43) | 23.82 (14.64)
  Mid Osteo cortical VOI BMD: number analyzed (Participants) | 42 | 50 | 43 | 43 | 41 | 49 | 36
  Mid Osteo cortical VOI BMD | -0.30 (4.69) | 0.63 (4.80) | 2.37 (6.37) | 2.57 (5.14) | 1.22 (4.39) | 4.98 (4.63) | 9.25 (7.68)

13. Secondary Outcome: Percent Change From Baseline to Month 12 in the Total Vertebra Integral VOI at the Lumbar Spine as Measured by QCT Scans
Description: QCT is a three-dimensional non-projectional technique to quantify BMD with a number of advantages to other densitometric techniques. Cortical and trabecular bone can be separated, trabecular VOI are largely independent of degenerative changes in the spine and 3 dimensional geometric parameters can be determined. BMD as measured by QCT is a true density measured in g/cm^3 in contrast to DXA Which determines an areal density measured in g/cm^2. Baseline values were assessed on Day 0. Percent change from Baseline was computed as (change from baseline / baseline value) * 100%.
Time Frame: Baseline (Day 0) and Month 12
Population: Intent-to-Treat population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change in VOI
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 42 | 50 | 43 | 43 | 41 | 49 | 36
Percent change in VOI | 0.04 (4.19) | 0.85 (4.14) | 3.01 (5.18) | 3.58 (5.70) | 3.54 (5.64) | 5.39 (5.87) | 12.23 (8.43)

14. Secondary Outcome: Percent Change From Baseline to Month 12 in the Volumetric Integral, Cortical, and Trabecular Density (BMD) at the Hip as Measured by QCT Scans
Description: QCT is a three-dimensional non-projectional technique to quantify BMD with a number of advantages to other densitometric techniques. Cortical and trabecular bone can be separated, trabecular VOI are largely independent of degenerative changes in the spine and 3 dimensional geometric parameters can be determined. BMD as measured by QCT is a true density measured in mg/cm^3 in contrast to DXA Which determines an areal density measured in g/cm^2. Baseline values were assessed on Day 0. Percent change from Baseline was computed as (change from baseline / baseline value) * 100%.
Time Frame: Baseline (Day 0) and Month 12
Population: Intent-to-Treat population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change in BMD
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 41 | 47 | 40 | 39 | 37 | 45 | 26
Percent change in BMD
  Femur integral VOI BMD | 0.02 (2.78) | -0.05 (2.67) | -0.81 (2.80) | -0.53 (2.18) | -0.15 (2.98) | 2.70 (2.13) | 3.92 (2.67)
  Femur trabecular VOI BMD | -0.36 (5.53) | -0.40 (6.81) | -2.16 (7.39) | 1.16 (5.06) | 2.81 (8.20) | 3.05 (5.92) | 13.19 (8.96)
  Femur cortical VOI BMD | 1.11 (4.04) | -0.32 (2.90) | -1.46 (2.81) | -1.06 (2.53) | -1.79 (3.01) | 2.44 (3.13) | 0.22 (2.63)
  Neck integral VOI BMD | -0.10 (2.48) | 0.16 (2.83) | -0.94 (3.34) | -1.20 (2.99) | -1.45 (3.22) | 1.65 (2.72) | 2.06 (3.65)
  Neck trabecular VOI BMD | -0.95 (7.44) | -2.19 (7.91) | -2.68 (6.14) | 1.35 (9.91) | 3.05 (11.18) | 2.77 (7.55) | 11.27 (10.31)
  Neck cortical VOI BMD | 1.23 (4.55) | 0.44 (4.16) | -1.67 (3.95) | -1.85 (3.89) | -2.80 (4.55) | 1.10 (4.25) | -0.69 (4.49)
  Trochanter integral VOI BMD | -0.58 (3.88) | -0.16 (4.22) | -1.53 (3.92) | -1.16 (3.29) | -0.98 (3.83) | 3.15 (3.27) | 4.96 (4.74)
  Trochanter trabecular VOI BMD | -1.62 (9.67) | -1.34 (13.50) | -2.54 (11.05) | 2.12 (8.82) | 2.10 (10.66) | 3.55 (7.55) | 14.12 (14.51)
  Trochanter cortical VOI BMD | 0.56 (5.29) | -0.70 (4.08) | -1.53 (3.60) | -1.48 (3.53) | -2.59 (4.04) | 3.33 (3.57) | 1.99 (4.37)

15. Secondary Outcome: Percent Change From Baseline to Month 12 in Cortical Thickness at the Hip as Measured by QCT Scans
Description: Percent change in thickness of femur neck cortical VOI thickness and trochanter cortical VOI thickness were at Month 12 measured by QCT were reported. Assessments performed on Day 0 were considered as Baseline. Percent change from Baseline was computed as (change from baseline / baseline value) * 100%.
Time Frame: Baseline (Day 0) and Month 12
Population: Intent-to-Treat population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change in cortical thickness
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 41 | 47 | 40 | 39 | 37 | 45 | 26
Percent change in cortical thickness
  Neck cortical VOI Thickness | -0.85 (7.09) | -0.13 (5.98) | 1.12 (5.75) | -0.88 (4.73) | 0.32 (4.93) | -0.13 (5.98) | 0.39 (4.36)
  Trochanter cortical VOI Thickness | -1.00 (5.85) | 0.76 (4.40) | 1.01 (5.15) | -0.82 (3.65) | 1.60 (3.70) | 0.81 (5.39) | 0.76 (2.93)

16. Secondary Outcome: Biochemical Markers of Bone Turnover: Levels of C-terminal Telopeptide α1 Chain of Type 1 Collagen (CTX1)
Description: Blood samples were collected at Baseline (Day 0), Week 4, Month 3, 6, and 12 for measurement of CTX1.
Time Frame: Baseline (Day 0), Week 4, Month 3, 6, and 12
Population: Intent-to-Treat population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: nanogram per litre (ng/L)
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41
nanogram per litre (ng/L)
  Baseline: number analyzed (Participants) | 88 | 82 | 81 | 87 | 84 | 87 | 41
  Baseline | 625.2 (1.05) | 635.3 (1.05) | 632.0 (1.05) | 587.9 (1.05) | 645.5 (1.05) | 630.4 (1.05) | 564.0 (1.07)
  Baseline, Placebo contrast: number analyzed (Participants) | 0 | 82 | 81 | 87 | 84 | 87 | 41
  Baseline, Placebo contrast |  | 1.02 (1.07) | 1.01 (1.07) | 0.94 (1.07) | 1.03 (1.07) | 1.01 (1.07) | 0.90 (1.09)
  Week 4: number analyzed (Participants) | 76 | 78 | 76 | 83 | 78 | 63 | 38
  Week 4 | 530.7 (1.05) | 515.2 (1.05) | 525.4 (1.05) | 506.1 (1.05) | 529.2 (1.05) | 288.0 (1.06) | 576.1 (1.08)
  Week 4, Placebo contrast: number analyzed (Participants) | 0 | 78 | 76 | 83 | 78 | 63 | 38
  Week 4, Placebo contrast |  | 0.97 (1.08) | 0.99 (1.08) | 0.95 (1.08) | 1.00 (1.08) | 0.54 (1.08) | 1.09 (1.10)
  Month 3: number analyzed (Participants) | 76 | 73 | 71 | 75 | 72 | 49 | 40
  Month 3 | 523.5 (1.05) | 598.5 (1.06) | 688.9 (1.06) | 723.2 (1.05) | 818.9 (1.06) | 257.1 (1.06) | 864.1 (1.08)
  Month 3, Placebo contrast: number analyzed (Participants) | 0 | 73 | 71 | 75 | 72 | 49 | 40
  Month 3, Placebo contrast |  | 1.14 (1.08) | 1.32 (1.08) | 1.38 (1.08) | 1.56 (1.08) | 0.49 (1.08) | 1.65 (1.10)
  Month 6: number analyzed (Participants) | 69 | 70 | 66 | 73 | 70 | 34 | 37
  Month 6 | 517.6 (1.06) | 648.2 (1.06) | 777.1 (1.06) | 859.6 (1.06) | 964.3 (1.06) | 235.9 (1.07) | 1112 (1.08)
  Month 6, Placebo contrast: number analyzed (Participants) | 0 | 70 | 66 | 73 | 70 | 34 | 37
  Month 6, Placebo contrast |  | 1.25 (1.08) | 1.50 (1.08) | 1.66 (1.08) | 1.86 (1.08) | 0.46 (1.09) | 2.15 (1.10)
  Month 12: number analyzed (Participants) | 50 | 44 | 49 | 40 | 49 | 50 | 37
  Month 12 | 525.1 (1.08) | 695.2 (1.08) | 806.1 (1.08) | 852.8 (1.08) | 991.9 (1.08) | 158.3 (1.08) | 1071 (1.10)
  Month 12, Placebo contrast: number analyzed (Participants) | 0 | 44 | 49 | 40 | 49 | 50 | 37
  Month 12, Placebo contrast |  | 1.32 (1.12) | 1.54 (1.11) | 1.62 (1.12) | 1.89 (1.11) | 0.30 (1.11) | 2.04 (1.13)

17. Secondary Outcome: Biochemical Markers of Bone Turnover: Procollagen Type 1 N-terminal Propeptide (P1NP)
Description: Blood samples were collected at Baseline (Day 0), Week 4, Month 3, 6, and 12 for measurement of P1NP.
Time Frame: Baseline (Day 0), Week 4, Month 3, 6, and 12
Population: Intent to treat population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Microgram per Litre (mcg/L)
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41
Microgram per Litre (mcg/L)
  Baseline: number analyzed (Participants) | 86 | 83 | 81 | 87 | 83 | 88 | 41
  Baseline | 47.66 (1.05) | 45.59 (1.05) | 47.70 (1.05) | 46.62 (1.05) | 46.19 (1.05) | 47.71 (1.05) | 48.57 (1.07)
  Baseline, Placebo contrast: number analyzed (Participants) | 0 | 83 | 81 | 87 | 83 | 88 | 41
  Baseline, Placebo contrast |  | 0.96 (1.07) | 1.00 (1.07) | 0.98 (1.07) | 0.97 (1.07) | 1.00 (1.07) | 1.02 (1.08)
  Week 4: number analyzed (Participants) | 80 | 78 | 75 | 85 | 79 | 81 | 39
  Week 4 | 45.32 (1.05) | 49.67 (1.05) | 57.36 (1.05) | 60.27 (1.05) | 63.46 (1.05) | 43.66 (1.05) | 92.74 (1.07)
  Week 4, Placebo contrast: number analyzed (Participants) | 0 | 78 | 75 | 85 | 79 | 81 | 39
  Week 4, Placebo contrast |  | 1.10 (1.07) | 1.27 (1.07) | 1.33 (1.07) | 1.40 (1.07) | 0.96 (1.07) | 2.05 (1.09)
  Month 3: number analyzed (Participants) | 77 | 72 | 72 | 76 | 73 | 79 | 40
  Month 3 | 39.53 (1.05) | 49.99 (1.05) | 65.21 (1.05) | 73.68 (1.05) | 86.84 (1.05) | 20.15 (1.05) | 99.74 (1.08)
  Month 3, Placebo contrast: number analyzed (Participants) | 0 | 72 | 72 | 76 | 73 | 79 | 40
  Month 3, Placebo contrast |  | 1.26 (1.08) | 1.65 (1.08) | 1.86 (1.08) | 2.20 (1.08) | 0.51 (1.07) | 2.52 (1.09)
  Month 6: number analyzed (Participants) | 69 | 70 | 67 | 72 | 70 | 74 | 38
  Month 6 | 38.41 (1.05) | 56.37 (1.05) | 75.73 (1.06) | 90.55 (1.05) | 104.6 (1.05) | 16.41 (1.05) | 117.8 (1.08)
  Month 6, Placebo contrast: number analyzed (Participants) | 0 | 70 | 67 | 72 | 70 | 74 | 38
  Month 6, Placebo contrast |  | 1.47 (1.08) | 1.97 (1.08) | 2.36 (1.08) | 2.72 (1.08) | 0.43 (1.08) | 3.07 (1.09)
  Month 12: number analyzed (Participants) | 50 | 44 | 50 | 40 | 49 | 51 | 37
  Month 12 | 40.74 (1.05) | 61.43 (1.05) | 82.69 (1.05) | 98.04 (1.05) | 112.6 (1.05) | 16.98 (1.05) | 119.0 (1.07)
  Month 12, Placebo contrast: number analyzed (Participants) | 0 | 44 | 50 | 40 | 49 | 51 | 37
  Month 12, Placebo contrast |  | 1.51 (1.08) | 2.03 (1.08) | 2.41 (1.08) | 2.76 (1.08) | 0.42 (1.08) | 2.92 (1.09)

18. Secondary Outcome: Biochemical Markers of Bone Turnover: Bone Specific Alkaline Phosphatase (BALP)
Description: Blood samples were collected at Baseline (Day 0), Week 4, Month 3, 6, and 12 for measurement of BALP.
Time Frame: Baseline (Day 0), Week 4, Month 3, 6, and 12
Population: Intent-to-Treat population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mcg/L
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
Number analyzed (Participants) | 90 | 87 | 82 | 88 | 87 | 89 | 41
mcg/L
  Baseline: number analyzed (Participants) | 89 | 84 | 81 | 88 | 86 | 89 | 41
  Baseline | 14.46 (1.04) | 14.96 (1.04) | 14.24 (1.04) | 15.06 (1.04) | 14.12 (1.04) | 14.31 (1.04) | 14.50 (1.05)
  Baseline, Placebo contrast: number analyzed (Participants) | 0 | 84 | 81 | 88 | 86 | 89 | 41
  Baseline, Placebo contrast |  | 1.03 (1.05) | 0.98 (1.05) | 1.04 (1.05) | 0.98 (1.05) | 0.99 (1.05) | 1.00 (1.07)
  Week 4: number analyzed (Participants) | 79 | 79 | 76 | 85 | 79 | 83 | 39
  Week 4 | 14.02 (1.04) | 14.72 (1.04) | 14.51 (1.04) | 15.97 (1.04) | 15.72 (1.04) | 13.68 (1.04) | 16.19 (1.06)
  Week 4, Placebo contrast: number analyzed (Participants) | 0 | 79 | 76 | 85 | 79 | 83 | 39
  Week 4, Placebo contrast |  | 1.05 (1.05) | 1.03 (1.06) | 1.14 (1.05) | 1.12 (1.05) | 0.98 (1.05) | 1.15 (1.07)
  Month 3: number analyzed (Participants) | 77 | 73 | 71 | 75 | 73 | 78 | 40
  Month 3 | 12.66 (1.04) | 15.23 (1.04) | 15.44 (1.04) | 18.77 (1.04) | 17.85 (1.04) | 9.44 (1.04) | 16.53 (1.06)
  Month 3, Placebo contrast: number analyzed (Participants) | 0 | 73 | 71 | 75 | 73 | 78 | 40
  Month 3, Placebo contrast |  | 1.20 (1.06) | 1.22 (1.06) | 1.48 (1.06) | 1.41 (1.06) | 0.75 (1.06) | 1.31 (1.07)
  Month 6: number analyzed (Participants) | 69 | 71 | 67 | 73 | 70 | 74 | 37
  Month 6 | 12.81 (1.04) | 16.31 (1.04) | 17.43 (1.04) | 22.18 (1.04) | 21.47 (1.04) | 8.36 (1.04) | 17.63 (1.06)
  Month 6, Placebo contrast: number analyzed (Participants) | 0 | 71 | 67 | 73 | 70 | 74 | 37
  Month 6, Placebo contrast |  | 1.27 (1.06) | 1.36 (1.06) | 1.73 (1.06) | 1.68 (1.06) | 0.65 (1.06) | 1.38 (1.07)
  Month 12: number analyzed (Participants) | 50 | 44 | 50 | 40 | 48 | 50 | 37
  Month 12 | 13.25 (1.04) | 16.64 (1.04) | 18.80 (1.04) | 23.36 (1.04) | 23.28 (1.04) | 8.42 (1.04) | 19.08 (1.06)
  Month 12, Placebo contrast: number analyzed (Participants) | 0 | 44 | 50 | 40 | 48 | 50 | 37
  Month 12, Placebo contrast |  | 1.26 (1.06) | 1.42 (1.06) | 1.76 (1.06) | 1.76 (1.06) | 0.64 (1.06) | 1.44 (1.07)

19. Secondary Outcome: Blood Concentrations of Ronacaleret
Description: Blood samples were collected and analyzed for concentrations of ronacaleret. The individual blood concentration-time data from the intensive PK-PD subgroup of participants were analyzed by standard noncompartmental methods. Blood concentrations of ronacaleret were reported.
Time Frame: Pre-dose (0.0 hour [h]) and 12 h post dose at Week 4, 20, 40 min, 1, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 1-4, 8-12, and 24 h at Month 3, 6 and 12
Population: Pharmacokinetic Concentration Population comprised of any Intent-to-Treat participants for whom a SB-751689 pharmacokinetic blood sample was obtained and analyzed. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD
Number analyzed (Participants) | 76 | 74 | 80 | 78
nanograms per millilitre (ng/mL)
  Week 4, Pre-dose: number analyzed (Participants) | 67 | 65 | 73 | 71
  Week 4, Pre-dose | 41.22 (127.438) | 37.24 (36.203) | 85.44 (158.849) | 79.40 (74.083)
  Week 4, 8-12 h post dose: number analyzed (Participants) | 66 | 64 | 72 | 70
  Week 4, 8-12 h post dose | 204.82 (183.245) | 328.33 (222.061) | 581.08 (360.031) | 685.14 (450.467)
  Month 6, Pre-dose: number analyzed (Participants) | 66 | 61 | 70 | 67
  Month 6, Pre-dose | 21.37 (19.769) | 65.94 (214.325) | 74.12 (146.094) | 117.94 (288.413)
  Month 6, 1-4 h post dose: number analyzed (Participants) | 49 | 45 | 51 | 53
  Month 6, 1-4 h post dose | 644.90 (408.282) | 1308.35 (943.397) | 1610.74 (1016.608) | 2054.71 (1499.079)
  Month 6, 8-12 h post dose: number analyzed (Participants) | 52 | 45 | 53 | 54
  Month 6, 8-12 h post dose | 186.69 (101.326) | 385.03 (284.963) | 576.35 (382.494) | 796.99 (640.016)
  Month 6, 24 h post dose: number analyzed (Participants) | 13 | 14 | 14 | 11
  Month 6, 24 h post dose | 186.21 (151.855) | 290.74 (125.486) | 578.63 (398.915) | 473.41 (237.671)
  Month 12, Pre-dose: number analyzed (Participants) | 43 | 43 | 38 | 42
  Month 12, Pre-dose | 20.68 (15.971) | 33.47 (26.747) | 147.63 (370.860) | 114.83 (179.448)
  Month 12, 1-4 h post dose: number analyzed (Participants) | 28 | 28 | 28 | 31
  Month 12, 1-4 h post dose | 779.92 (465.356) | 999.63 (659.880) | 1819.53 (1021.984) | 2128.24 (1549.003)
  Month 12, 8-12 h post dose: number analyzed (Participants) | 30 | 28 | 27 | 30
  Month 12, 8-12 h post dose | 203.39 (124.866) | 262.20 (137.152) | 651.95 (391.752) | 740.18 (679.348)
  Month 12, 24 h post dose: number analyzed (Participants) | 12 | 14 | 9 | 11
  Month 12, 24 h post dose | 187.23 (100.001) | 297.20 (146.806) | 626.72 (231.777) | 512.65 (314.692)

20. Secondary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUC 0-t) and Area Under the Concentration-time Curve Over the Dosing Interval (AUC 0-tau) of Ronacaleret
Description: Blood samples were collected and analyzed for concentrations of ronacaleret. The individual blood concentration-time data from the intensive pharmacokinetic and pharmacodynamics subgroup of participants were analyzed by standard noncompartmental methods. Blood samples were collected and analyzed for concentrations of ronacaleret. The individual blood concentration-time data from the intensive PK-PD subgroup of participants were analyzed by standard noncompartmental methods. Following log transformation, AUC(0-t) and AUC(0-τ) of ronacaleret were separately analyzed by ANOVA using mixed effects model, fitting treatment and country/region as fixed effects.
Time Frame: Pre-dose (0.0 h) and 12 h post dose at Week 4, 20, 40 min, 1, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 1-4, 8-12, and 24 h at Month 3, 6 and 12
Population: Pharmacokinetic Parameters Population comprised of any participant in the pharmacokinetic concentration population who provided pharmacokinetic parameters. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per millilitre (ng*hr/mL)
Arm/Group | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD
Number analyzed (Participants) | 13 | 14 | 14 | 11
nanogram*hour per millilitre (ng*hr/mL)
  AUC 0-t, Month 6 | 2495.8751 (53.13) | 4575.8746 (35.50) | 7545.3302 (42.26) | 6712.0537 (79.69)
  AUC 0-t, Month 12: number analyzed (Participants) | 12 | 14 | 9 | 11
  AUC 0-t, Month 12 | 2766.6822 (64.20) | 4548.6490 (43.87) | 9259.3127 (37.74) | 6798.4219 (65.17)
  AUC 0-tau, Month 6 | 3628.0901 (66.72) | 6428.5540 (36.62) | 10825.9083 (50.48) | 9810.4614 (80.08)
  AUC 0-tau, Month 12: number analyzed (Participants) | 12 | 14 | 9 | 11
  AUC 0-tau, Month 12 | 3922.9369 (75.72) | 6455.1756 (42.03) | 14827.6940 (38.28) | 10079.2847 (71.01)

21. Secondary Outcome: Maximum Blood Concentration (Cmax) of Ronacaleret
Description: Blood samples were collected and analyzed for concentrations of ronacaleret. The individual blood concentration-time data from the intensive pharmacokinetic and pharmacodynamics subgroup of participants were analyzed by standard noncompartmental methods. Blood samples were collected and analyzed for concentrations of ronacaleret. The individual blood concentration-time data from the intensive PK-PD subgroup of participants were analyzed by standard noncompartmental methods. Following log transformation, Cmax of ronacaleret were separately analyzed by ANOVA using mixed effects model, fitting treatment and country/region as fixed effects.
Time Frame: as for outcome 20
Population: Pharmacokinetic parameter population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD
Number analyzed (Participants) | 13 | 14 | 14 | 11
ng/mL
  Cmax. Month 6 | 572.10 (44.79) | 1050.42 (40.82) | 1756.45 (52.80) | 1556.58 (76.83)
  Cmax. Month 12: number analyzed (Participants) | 12 | 14 | 9 | 11
  Cmax. Month 12 | 661.70 (74.39) | 999.91 (37.18) | 2254.26 (41.57) | 1506.45 (63.78)

22. Secondary Outcome: Time Required to Achieve Maximum Concentration of Ronacaleret in Blood (Tmax)
Description: Blood samples were collected and analyzed for concentrations of ronacaleret. The individual blood concentration-time data from the intensive pharmacokinetic and pharmacodynamics subgroup of participants were analyzed by standard noncompartmental methods.
Time Frame: as for outcome 20
Population: Pharmacokinetic parameters population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD
Number analyzed (Participants) | 13 | 14 | 14 | 11
h
  Tmax, Month 6 | 1.483 [0.98 to 4.02] | 1.250 [0.67 to 3.03] | 1.700 [0.33 to 3.02] | 1.500 [0.67 to 4.07]
  Tmax, Month 12: number analyzed (Participants) | 12 | 14 | 9 | 11
  Tmax, Month 12 | 1.000 [0.33 to 4.00] | 1.500 [0.67 to 2.95] | 1.500 [0.00 to 2.58] | 1.500 [0.33 to 3.00]

ADVERSE EVENTS:
Time Frame: Up to Follow-up visit (12 month and 2 weeks)
Description: Intent-to-Treat population was used to report AEs
Arm/Group | Placebo | Ronacaleret, 100 mg Tablet, OD | Ronacaleret, 200 mg Tablet, OD | Ronacaleret, 300 mg Tablet, OD | Ronacaleret, 400 mg Tablet, OD | Alendronate, 70 mg, Capsule, OW | Teriparatide, 20 mcg, SC Injection, OD
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/87 | 0/82 | 0/88 | 0/87 | 0/89 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/90 | 2/87 | 5/82 | 7/88 | 3/87 | 6/89 | 4/41
Other Adverse Events (participants affected / at risk) | 54/90 | 54/87 | 57/82 | 55/88 | 61/87 | 46/89 | 30/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=90) | Ronacaleret, 100 mg Tablet, OD (N=87) | Ronacaleret, 200 mg Tablet, OD (N=82) | Ronacaleret, 300 mg Tablet, OD (N=88) | Ronacaleret, 400 mg Tablet, OD (N=87) | Alendronate, 70 mg, Capsule, OW (N=89) | Teriparatide, 20 mcg, SC Injection, OD (N=41)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperplasia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Smear cervix abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salpingo-oophorectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=90) | Ronacaleret, 100 mg Tablet, OD (N=87) | Ronacaleret, 200 mg Tablet, OD (N=82) | Ronacaleret, 300 mg Tablet, OD (N=88) | Ronacaleret, 400 mg Tablet, OD (N=87) | Alendronate, 70 mg, Capsule, OW (N=89) | Teriparatide, 20 mcg, SC Injection, OD (N=41)
Nasopharyngitis (Infections and infestations) | 17 | 16 | 13 | 12 | 16 | 12 | 7
Influenza (Infections and infestations) | 7 | 6 | 5 | 6 | 9 | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 5 | 4 | 2 | 8 | 3 | 2
Bronchitis (Infections and infestations) | 5 | 4 | 3 | 4 | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 4 | 6 | 0 | 3 | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 5 | 0 | 1 | 2 | 2 | 4
Tooth infection (Infections and infestations) | 1 | 2 | 0 | 4 | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 8 | 11 | 12 | 5 | 1
Nausea (Gastrointestinal disorders) | 4 | 1 | 6 | 9 | 11 | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 6 | 3 | 6 | 3 | 4 | 3
Constipation (Gastrointestinal disorders) | 2 | 5 | 4 | 9 | 5 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 3 | 6 | 4 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 5 | 0 | 3 | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7 | 9 | 5 | 10 | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 6 | 2 | 6 | 6 | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 0 | 4 | 3 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 2 | 1 | 0 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 1 | 1 | 5 | 0
Headache (Nervous system disorders) | 7 | 5 | 5 | 4 | 4 | 8 | 6
Dizziness (Nervous system disorders) | 4 | 5 | 8 | 5 | 10 | 0 | 6
Hypertension (Vascular disorders) | 4 | 5 | 5 | 2 | 3 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 3 | 2 | 2 | 2 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 4 | 2 | 1 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 2 | 5 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated for futility in a phased manner by the sponsor on 25-Sep-2008 once the results of a planned 6-month interim analysis were available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.